CLINICAL TRIAL: NCT05269251
Title: Effects of Brachial Plexus Block Applied With Different Approaches on Tissue Oxygenation
Brief Title: Effects of Brachial Plexus Block on Tissue Oxygenation
Acronym: BrachialPlexus
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Demet Coşkun, Associate Professor M.D, Gazi University
Other Study IDs: 357
Record Dates: First submitted 2022-02-25; First posted 2022-03-07 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Tissue Oxygenation
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Axillary Brachial Plexus Block: Our study includes 3 groups, 33 patients each who underwent axillary, infraclavicular and interscalene blocks. In the study, which of the axillary, infraclavicular and interscalene blocks will be preferred, will be decided by an experienced anesthesiologist in accordance with the type of surgery to be performed. Demographic data, comorbidities, and smoking will be questioned in each group, arterial blood pressure, heart rate, body temperature, radial artery diameter and flow velocities will be recorded before peripheral nerve block is applied, and tissue oxygenation will be measured with Near Infrared Spectroscopy (NIRS) in the extremities with and without block. Tissue oxygenation, radial artery flow velocity and diameters, body temperature will be measured simultaneously at 0(basal)-5-10-15-20-25 and 30th minutes after the application of the block. test will be applied and the success of the procedure will be determined accordingly.
  Interventions: Device: Near Infrared Spectroscopy (NIRS)
- Infraclavicular Brachial Plexus Block: Our study includes 3 groups, 33 patients each who underwent axillary, infraclavicular and interscalene blocks. In the study, which of the axillary, infraclavicular and interscalene blocks will be preferred, will be decided by an experienced anesthesiologist in accordance with the type of surgery to be performed. Demographic data, comorbidities, and smoking will be questioned in each group, arterial blood pressure, heart rate, body temperature, radial artery diameter and flow velocities will be recorded before peripheral nerve block is applied, and tissue oxygenation will be measured with Near Infrared Spectroscopy (NIRS) in the extremities with and without block. Tissue oxygenation, radial artery flow velocity and diameters, body temperature will be measured simultaneously at 0(basal)-5-10-15-20-25 and 30th minutes after the application of the block. test will be applied and the success of the procedure will be determined accordingly.
  Interventions: Device: Near Infrared Spectroscopy (NIRS)
- Interscalene Brachial Plexus Block: Our study includes 3 groups, 33 patients each who underwent axillary, infraclavicular and interscalene blocks. In the study, which of the axillary, infraclavicular and interscalene blocks will be preferred, will be decided by an experienced anesthesiologist in accordance with the type of surgery to be performed. Demographic data, comorbidities, and smoking will be questioned in each group, arterial blood pressure, heart rate, body temperature, radial artery diameter and flow velocities will be recorded before peripheral nerve block is applied, and tissue oxygenation will be measured with Near Infrared Spectroscopy (NIRS) in the extremities with and without block. Tissue oxygenation, radial artery flow velocity and diameters, body temperature will be measured simultaneously at 0(basal)-5-10-15-20-25 and 30th minutes after the application of the block. test will be applied and the success of the procedure will be determined accordingly.
  Interventions: Device: Near Infrared Spectroscopy (NIRS)

INTERVENTIONS:
Device: Near Infrared Spectroscopy (NIRS) — After the brachial plexus block, the regional oxygen saturation (rSO2) was monitored for 30 minutes with the Regional Oximetry System (O3™, Masimo, Irvine, CA) and the radial artery diameter with ultrasound in the same period.
  Other Names: Regional Oximetry System (O3™, Masimo, Irvine, CA)

SUMMARY:
The aim of this study is to measure the effects of sympathetic blockade caused by peripheral nerve blocks performed with the axillary, infraclavicular and interscalene approach on tissue oxygenation with Near Infrared Spectroscopy (NIRS), to evaluate and compare the radial artery flow velocity and diameter in the blocked extremity, and to investigate whether there is a relationship with the quality of the sensory and motor block.

DETAILED DESCRIPTION:
It has been reported that vasodilation after peripheral nerve blocks increases tissue oxygenation and increases arterial circulation on the ipsilateral side . Near Infrared Spectroscopy (NIRS), a noninvasive measurement method of tissue oxygen level, is used to measure regional hemoglobin oxygen saturation of arterial, venous and capillary blood .

Many studies have compared the effects of upper extremity peripheral nerve blocks on the onset, quality, extent, and postoperative pain of sensory and motor block through axillary, infraclavicular, supraclavicular and interscalene approaches.

The aim of this study is to measure the effects of sympathetic blockade caused by peripheral nerve blocks performed with the axillary, infraclavicular and interscalene approach on tissue oxygenation with Near Infrared Spectroscopy (NIRS), to evaluate and compare the radial artery flow velocity and diameter in the blocked extremity, and to investigate whether there is a relationship with the quality of the sensory and motor block.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients
* Patients between the ages of 18 and 65
* Patients who applied axillary block
* Patients who applied infraclavicular block
* Patients who applied interscalene block

Exclusion Criteria:

* Peripheral nerve disease a history
* History of thrombosis in the extremity to be blocked
* History of embolism in the extremity to be blocked
* Presence of neuropathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ASA I-III patients aged 18-65 years, who were decided to apply axillary,infraclavicular and interscalene blocks as the anesthesia method, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
tissue oxygenation | 30 minutes
  Measured from both extremities by Near Infrared Spectroscopy for 30 min after brachial nerve block.

SECONDARY OUTCOMES:
Radial artery diameter | 30 minutes
  measured on the side of the block after brachial nerve block

CONTACTS AND LOCATIONS:
Locations (1):
- Demet Coskun, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No